CLINICAL TRIAL: NCT01751737
Title: Investigation of the Magnitude of Uptake, Retention, and Spatial Distribution Pattern of 18F-Choline in Comparison With MRI and Histology Obtained From Prostate Cancer Biopsies
Brief Title: Choline PET/CT and MRI for Targeted Prostate Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Morand Piert, MD, Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00059514
Record Dates: First submitted 2012-11-30; First posted 2012-12-18 (Estimated); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Prostate Cancer
Keywords: prostate; cancer; biopsy; 18F-choline; PET; MRI
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prostate Cancer Imaging (Experimental): Subjects will receive multi-sequence Magnetic Resonance Imaging (MRI) of the prostate and pelvis. This scan will take approximately 90 minutes.
  In addition, a 18F-Choline PET/CT(Positron emission tomography/computed tomography) scan of the abdomen and pelvis is performed. This scan will take about 30 minutes. Subjects may receive an additional 30 minute scan, if needed.
  Patients participating in an active surveillance program at the University of Michigan may receive yearly imaging followed by a prostate biopsy procedure.
  Interventions: Procedure: Prostate Cancer Imaging

INTERVENTIONS:
Procedure: Prostate Cancer Imaging — After imaging is completed, subjects will be scheduled for a prostate biopsy performed as part of their clinical care. If the imaging has identified suspicious lesions in the prostate, these regions will be made visible for the Urologist to be targeted for additional biopsies. These additional biopsies will undergo histological evaluation and further metabolomic testing to better understand metabolic differences between various grades of prostate cancer lesions.

SUMMARY:
This research study will access the using of a radiotracer, 18F-choline PET/CT and MRI for prostate cancer in patients undergoing diagnostic prostate biopsy. Patients receive MRI guided prostate biopsies and metabolomic profiling of prostate biopsy tissues.

DETAILED DESCRIPTION:
This is an explorative diagnostic basic research study to assess the value of 18F-choline PET/CT and multi-sequence MRI for prostate cancer in patients undergoing diagnostic prostate biopsy. Patients will receive image-guided (targeted) prostate biopsies and metabolomic profiling of prostate biopsy tissues to evaluate underlying metabolic changes in comparison with pathological Gleason grading.

ELIGIBILITY:
Inclusion Criteria:

* Males 40 years of age or older scheduled for prostate biopsy (for known or suspected prostate cancer) followed by planned prostatectomy (population group A)
* Males 40 years of age or older with known (biopsy-confirmed) primary adenocarcinoma of the prostate undergoing active surveillance scheduled for prostate biopsy (population group B)

Exclusion Criteria:

* Androgen ablation (hormone treatment) within the last 3 months
* Prostate biopsy within 6 weeks prior to PET or MRI imaging
* Active inflammatory bowel disease within the last 6 months
* Acute prostatitis within the last 6 months
* A non-urologic bacterial infection requiring active treatment with antibiotics
* Active other malignancy (except basal cell or squamous cell skin cancer) within the last 2 years
* Previous radiation treatment of the pelvis
* Symptomatic distal rectal stenosis
* Known hypersensitivity to glucagon
* Pheochromocytoma, insulinoma or galactosemia
* Insulin-dependent diabetes

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Evaluation whether the odds of primary Gleason ≥ 3+4 are greater for image-guided biopsy (based on parametric PET/MRI) than for non-image-guided (standard) biopsy. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Morand R. Piert, M.D., Principal Investigator — University of Michigan Hospital
Locations (1):
- University of Michigan Health Systems, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Piert M, Montgomery J, Kunju LP, Siddiqui J, Rogers V, Rajendiran T, Johnson TD, Shao X, Davenport MS. 18F-Choline PET/MRI: The Additional Value of PET for MRI-Guided Transrectal Prostate Biopsies. J Nucl Med. 2016 Jul;57(7):1065-70. doi: 10.2967/jnumed.115.170878. Epub 2016 Mar 16. PMID 26985061